CLINICAL TRIAL: NCT00811057
Title: Tocolysis for Preterm Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Rick Martin, Associate Professor Maternal-Fetal Medicine; Dept of Ob-Gyn, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0249
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-02

CONDITIONS: Preterm Labor
Keywords: Preterm Labor in Pregnancy
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Nifedipine; Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 Magnesium Sulfate (Active Comparator)
  Interventions: Drug: 1 Magnesium Sulfate
- 2 Nifedipine (Active Comparator): Participants randomized to this group will receive the medication nifedipine orally.
  Interventions: Drug: Nifedipine
- 3 Indomethacin (Active Comparator): Participants randomized to this arm will receive the medication indomethacin per rectum and orally.
  Interventions: Drug: Indomethacin

INTERVENTIONS:
Drug: 1 Magnesium Sulfate — Participants randomized to this arm will receive a loading dose of 6gms intravenously followed by a maintenance dose of 2-4gm/hr, per physician discretion, until uterine quiescence is achieved. The Magnesium Sulfate dosage is then titrated down until discontinued per physician discretion.
  Arms: 1 Magnesium Sulfate
Drug: Nifedipine — Participants randomized to receive nifedipine will receive an initial 30mg loading dose, then 10 - 20mg q 4 - 6 hours as needed, per physician discretion, until uterine quiescence is achieved.
  Arms: 2 Nifedipine
Drug: Indomethacin — Participants randomized to receive indomethacin will receive an initial 100mg per rectum X1, may repeat x1, and then 25 - 50mg orally every 6 hours over 48 hours as needed per physician discretion until uterine quiescence has been achieved.
  Arms: 3 Indomethacin

SUMMARY:
Preterm birth is the most common and costly complication in obstetrics. It complicates up to 11% of all pregnancies and it is responsible for 70% of sick babies. The ideal way to stop preterm labor when it occurs (which drug to use) is not known. Currently magnesium sulfate is used by about 95% of all practitioners, but recent data suggest magnesium given this way may be harmful for the baby's future development. Other drugs such as antiprostaglandin agents are very effective in stopping uterine activity, but particularly when used for >48 hours have been associated with both maternal and fetal sides effects. Lastly, calcium channel antagonists are effective in stopping contractions and have very little in the way of maternal and fetal side effects, but less data is available in the United States on their use. Because there is no FDA approved drug to stop preterm labor, we purpose to randomize all women with preterm labor (20-34 weeks) to receive one of the above three methods of stopping preterm labor. The primary outcomes will be to see which agent stops the uterine contractions most effectively, for the longest period of time with fewest relapses and results in significant prolongation of pregnancy. If one of these agents is clearly superior to the other two it would help women avoid early delivery or have significant extension of their pregnancy to avoid some of the complications of preterm birth in the baby.

DETAILED DESCRIPTION:
Preterm labor is the most common complication of pregnancy and one of the most catastrophic occurring in 10-12% of all pregnancies and accounting for up to 80% of the neonatal morbidity1. In addition, the delivery of a very low birth weight baby often leads to a reduction in cognitive and academic skills as well an increased in mental retardation by age five2,3. While there are many strategies to treat women in preterm labor all of the agents which have been used have side effects, acutely prolong the pregnancy only for a few days, and there have been no universally accepted treatment for long term prolongation using oral tocolytics in the home4,5,6. While beta-agonists have been used for several decades as primary agents for acute tocolysis, side effects have led to these agents being relegated to adjunctive therapy or in home care program with the programmable subcutaneous pump7. Consequently there are no tocolytic agents approved by the FDA for use during pregnancy.

The most common drug used for acute tocolysis is magnesium sulfate, which is administered intravenously to stop contractions8. While it appears to be effective for short-term tocolysis it is thought to be not as effective as anti-prostaglandins or calcium channel antagonists in quickly suppressing uterine activity. In addition, there has been controversy as to adverse effects on the neonate when this drug is used to impede uterine contractions9. Some authors feel that it causes adverse neurologic function in the baby where as others feel that it is not associated with any increase neonatal morbidity/mortality in premature infants9.10. Regardless, for clinicians treating women in preterm labor magnesium remains the main stay of therapy.

Newer developments, however, point to the improved effectiveness of anti-prostaglandin agents and calcium channel antagonists as it concerns treating such patients7,11. Calcium channel antagonists are just as effective and appear to be safer than magnesium for primary tocolytic treatment of women in preterm labor12-14. Tocolytic treatment with anti-prostaglandin drugs such as indomethacin, a Cox-1 inhibitor, has demonstrated them to be the most effective and most rapid tocolytic agent available15. Initially there were reports of increasing complications with the use of this drug16,17. However, it has been shown that these concerns are unwarranted if indomethacin use is limited to 48 hours per treatment cycle and the amniotic fluid assessed for oligohydramnios; therefore, in pregnancies <32 weeks there ample evidence to justify its use as a primary tocolytic18,19,20. This is particularly true with the newer agents of this class (Cox-2 inhibitors) which have fewer fetal side effects7,11. In sum, however, there are no randomized trials which demonstrate the effectiveness of these three types of agents.

B. Specific Aim

The purpose of this study is to compare the three categories of clinically used tocolytic agents in a prospective study that will allow direct comparison of outcomes in women with confirmed preterm labor. While magnesium sulfate tocolysis for acute treatment of preterm labor is the standard of care, there appear to be better tocolytic agents with less maternal and fetal side effects which could be used as primary agents.

C. Rationale

While there is no evidence that primary tocolytic agents such as magnesium sulfate or beta-agonist drugs prolong pregnancy extensively when compared to placebo, preterm labor and early delivery remain one of the top few health problems in the perinatal field. For that reason, investigations to compare available first line agents are warranted. Based on the current information in the literature calcium channel antagonists and anti-prostaglandin drugs are the best hope to treat acute preterm labor in an effort to significantly prolong pregnancy with the fewest adverse effects on mother and baby.

D. Benefit to Risk Ratio There is no tocolytic agent approved by the FDA and more importantly there is no drug used for this purpose that is free of maternal and fetal side effects. However, any treatment involves less risk than a preterm delivery. Because of long experience in the medical community, magnesium sulfate remains the number one choice of obstetricians throughout the United States, but it has a rather high rate of maternal side effects often leading to discontinuation of the drug. For acute treatment of preterm labor both calcium channel antagonists as well as anti-prostaglandins appear be more effective while having equal or better safety profiles for the mother and baby when used appropriately. The benefits of effectively prolonging pregnancy for several weeks far outweigh any medication effects to the mother or fetus and therefore, make continued investigation in these drugs reasonable.

E. Patient Population Patients will be recruited from the labor and delivery area of the University of Mississippi Medical Center. All patients who meet admission criteria will be offered participation in the study.

F. Materials and Methods

Patients who are experiencing confirmed preterm labor (regular uterine contractions, usually < 5 minutes apart, associated with cervical change such as dilatation and/or effacement) would be considered as potential participants.

After preterm labor has been confirmed and informed consent has been obtained, patients will be randomized by the use of sequentially numbered, sealed opaque envelopes to receive intravenous magnesium (6gm load plus 6gm/per hour IV to abolish contractions) versus a calcium channel antagonist (nifedipine 30mg loading, then 10 - 20mg q 4 - 6 hours) versus antiprostaglandin (indomethacin 100mg rectal suppositories may repeat x1 and then 25 - 50mg q 6 hours over 48 hours). The amount of each tocolytic over time will be recorded. If this fails to abolish uterine activity and there is no contraindication to continuing pregnancy (eg abruptio placenta, chorioamnionitis, non-reassuring fetal tracing, etc.) subcutaneous terbutaline (beta-agonist) will be given subcutaneously (250mg) as an adjunctive measure to abolish contractions. As is our routine we will use blood tests, amniotic fluid assessment and ultrasound to detect infection or abruptio placenta which would lead to delivery after cessation of tocolytic treatment.

If there is continued failure of tocolysis further treatment will rest with the physician although in most cases the pregnancy will be delivered by this time due to continued contractions or diagnosis of complications listed above which contraindicate the continuation of the gestation.

Women will be separately randomized dependent on cervical status (0 - 3cm versus 4 - 6cm dilatation) to the same three choices. All other hospital management such as corticosteroid therapy to promote fetal lung maturity, continuous fetal heart rate monitoring, amnioinfusion, etc., and will be same regardless of group assessment, as is our standard of care.

G. Data Analysis

Data analysis will be by standard statistical methodology.

VII. Number of Patients Needed:

A sample size estimation indicates that 240 patients (80 in each group) will be necessary to have an 80% power (decreasing deliveries at < 32 weeks by 50%) of detecting a significance of < 0.05 in the number of preterm births. Likewise, in the > 4cm group (assuming 90% delivery within seven days) 40 patients in each group (120 women) will be necessary to have an 80% power of detecting (with a 25% reduction in deliveries with seven days) a significance of < 0.05. It is anticipated that it will take a time period of approximately two years to enroll this number of participants.

VIII. Research Equipment Needed:

None

ELIGIBILITY:
Inclusion Criteria:

* Pregnancies with intact membranes in confirmed preterm labor;
* 20 - 32 weeks' gestation;
* Cervical dilatation 0 - 3cm versus 4 - 6cm;
* No conditions contraindicating continued pregnancy (severe IUGR, chorioamnionitis, non-reassuring fetal tracing - physician judgement); AND
* Able and willing to consent to the study protocol.

Exclusion Criteria:

* Failure to meet admission criteria;
* Known serious fetal malformations;
* Severe maternal/obstetric disease affecting the mother or fetus (severe cardiac disease, placental abruption/previa, severe diabetes, severe preeclampsia, etc. - physician judgment);
* Allergic to magnesium, antiprostaglandin or calcium channel antagonist;
* Refusal or inability to consent to the study

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 301 (Actual)
Dates: Start 2004-06; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rick W Martin, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- The Winfred L. Wiser Hospital for Women and Infants at the University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were hospitalized in labor and delivery at University of Mississippi Medical Center in active preterm labor.
Groups:
- 1 Magnesium Sulfate: 1 Magnesium Sulfate : Participants randomized to this arm will receive a loading dose of 6gms intravenously followed by a maintenance dose of 2-4gm/hr, per physician discretion, until uterine quiescence is achieved. The Magnesium Sulfate dosage is then titrated down until discontinued per physician discretion.
- 2 Nifedipine: Participants randomized to this group will receive the medication nifedipine orally.
  Nifedipine : Participants randomized to receive nifedipine will receive an initial 30mg loading dose, then 10 - 20mg q 4 - 6 hours as needed, per physician discretion, until uterine quiescence is achieved.
- 3 Indomethacin: Participants randomized to this arm will receive the medication indomethacin per rectum and orally.
  Indomethacin : Participants randomized to receive indomethacin will receive an initial 100mg per rectum X1, may repeat x1, and then 25 - 50mg orally every 6 hours over 48 hours as needed per physician discretion until uterine quiescence has been achieved.
Period: Overall Study
Arm/Group | 1 Magnesium Sulfate | 2 Nifedipine | 3 Indomethacin
Started | 90 | 114 | 97
Completed | 85 | 104 | 87
Not Completed | 5 | 10 | 10
Not completed — Protocol Violation | 5 | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Magnesium Sulfate | 2 Nifedipine | 3 Indomethacin | Total
Number analyzed (Participants) | 90 | 114 | 97 | 301
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 90 | 114 | 97 | 301
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 23.9 (5.4) | 22.2 (4.3) | 22.9 (4.8) | 22.5 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 114 | 97 | 301
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 90 | 114 | 97 | 301

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure of This Research is to Compare the Efficacy of the Three Clinically Used Tocolytic Agents in a Prospective Study That Will Allow Direct Comparison of Outcomes in Women With Confirmed Preterm Labor.
Description: Gestational age at delivery in weeks.
Time Frame: 3-5 days after delivery
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | 1 Magnesium Sulfate | 2 Nifedipine | 3 Indomethacin
Number analyzed (Participants) | 90 | 114 | 97
weeks | 31.2 (3.9) | 31.8 (4.5) | 31.8 (4.2)

2. Secondary Outcome: The Secondary Outcome Measure of This Research is the Days Gained After Treatment to Delivery
Description: Days gained after treatment to delivery
Time Frame: after delivery of the infant
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 1 Magnesium Sulfate | 2 Nifedipine | 3 Indomethacin
Number analyzed (Participants) | 90 | 114 | 97
days | 22.5 (43.8) | 21.7 (21.7) | 22.7 (21.1)

ADVERSE EVENTS:
Arm/Group | 1 Magnesium Sulfate | 2 Nifedipine | 3 Indomethacin
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/114 | 0/97
Other Adverse Events (participants affected / at risk) | 0/90 | 0/114 | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No